CLINICAL TRIAL: NCT00499200
Title: A Positron Emission Tomography Study to Assess the Level and Duration of Occupancy of Serotonin-1A Receptors Produced by Single Oral Doses of SRA-444 in Healthy Elderly Subjects and in Subjects With Alzheimer Disease
Brief Title: Study Evaluating Safety, Tolerability, Pharmacokinetics and 5 HT1A Receptor Occupancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3197A1-1104
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- SRA-444 + Placebo (Experimental): Experimental; Placebo
  Interventions: Drug: SRA-444

INTERVENTIONS:
Drug: SRA-444

SUMMARY:
The study will include a preliminary pharmacokinetics (PK) / safety / tolerability evaluation in healthy elderly subjects followed by the Receptor Occupancy (RO) evaluations in healthy elderly subjects and in Alzheimer's Disease (AD) subjects.

ELIGIBILITY:
Inclusion criteria:

* Men or women from 60 years of age at screening.
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG).

Exclusion criteria:

* History of drug abuse within 1 year before study day 1.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of ascending single oral doses of SRA-444 in healthy elderly subjects and subjects with Alzheimer's disease | after each dose group completion
To obtain PK profiles and determine the level and duration of 5-HT1A RO of SRA-444 by PET | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Sweden: MedInfoNord@wyeth.com
Locations (1):
- Uppsala, Sweden